CLINICAL TRIAL: NCT04732377
Title: Analgesic Efficacy of Dexmedetomidine as Adjuvant to Levobupivacaine in Ultrasound-guided Erector Spinae Plan Block for Modified Radical Mastectomy
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: South Egypt Cancer Institute (Other)
Responsible Party: Principal Investigator, Peter Rafaat Edward Iskander, specialist, South Egypt Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: peter 3 SECI
Record Dates: First submitted 2021-01-09; First posted 2021-02-01 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain | interventions — Bupivacaine; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP(A) (CONTROL GROUP) (Placebo Comparator): Patient will receive 20 ml 0.25% levobupivacaine into interfascial plane below erector spinae muscle at level of T5.
  Interventions: Procedure: erector spinae block with bupivacaine
- Group (D) (Active Comparator): Patient will receive 20ml 0.25% levobupivacaine above + 1μ/kg dexmedetomidine into interfascial plane below erector spinae muscle at level of T5.
  Interventions: Procedure: erector spinae block with bupivacaine and dexmedetomidine

INTERVENTIONS:
Procedure: erector spinae block with bupivacaine — Group (A) (control group):
  Patient will receive 20 ml 0.25% levobupivacaine into interfascial plane below erector spinae muscle at level of T5.
  Arms: GROUP(A) (CONTROL GROUP)
Procedure: erector spinae block with bupivacaine and dexmedetomidine — Patient will receive 20ml 0.25% levobupivacaine above + 1μ/kg dexmedetomidine into interfascial plane below erector spinae muscle at level of T5.
  Arms: Group (D)

SUMMARY:
To evaluate the analgesic efficacy of dexmedetomidine as adjuvants to levobupivacaine in erector spinae plane block in modified radical mastectomy surgery.

DETAILED DESCRIPTION:
Premedication will be given, after complete fasting hours after applying standard monitors (noninvasive blood pressure, pulse oximetery, ECG, temperature and capnography), an intravenous cannula will be placed and secured.

Ultrasound guided Erector spinae plane (ESP) block will be given with patient in sitting position depending on surgical site (left or right) ESP block will be given using high frequency linear u/s transducer, the probe is placed in longitudinal orientation lateral to thoracic fifth spinous process, then Trapezius muscle, Rhomboidus major muscle, and erector spinae muscle, are identified from surface, we deposite20 ml of 0.25% levobupivacaine into interfacial plane below erector spinae muscle.

General anesthesia will be induced with fentanyl l μg /kg, propofol 2mg /kg, muscle relaxant (atracurium 0.5 mg/kg) inhalational anesthesia (isoflurane or sevoflurane) No other narcotic, analgesic or sedative will be administrated during operative period.

Standard monitor (mean arterial blood pressure, heart rate , oxygen saturation & end-tidal Co2) will observed and recorded every 30 min till end of surgery

Post-operative:

The patient will be transferred to the post anesthesia care unit (PACU) and will be monitored for:

1. Vital signs (heart rate, noninvasive blood pressure, and oxygen saturation).
2. RASS score (Richmond Agitation & Sedation scale) with its +4:-5 score range will be used to assess sedation post-operative, considered sedation ≥-2 table (1)
3. Numerical Rating Score (NRS) pain score with its 0-10 score range will be used to assess pain immediately post-operative and then at 2, 4, 6, 8, 12,18and 24hour in the post-operative period figure (1). (4)Time and amount to request analgesia (PCA patient controlled analgesia morphine (demand dose 1-2 mg, lock out 6-10 min)) at NRS≥3. (5) Side effect of studied drugs as (hypotension, sedation , respiration depression and vomiting ) and complication of the block for 24h post- operative.

ELIGIBILITY:
Inclusion Criteria:

* female patient
* American society of anesthesiologists (ASA) I and II physical status
* age from 25 to 70 years old
* scheduled for either left or right modified radical mastectomy (MRM).

Exclusion Criteria:

* infection of the skin at or near site of needle puncture,
* coagulopathy,
* drug hypersensitivity or allergy to the studied drugs,
* central or peripheral neuropathy,
* significant organ dysfunction cardiac dysrrhythmias,
* obesity (BMI>35kg/m2)
* recently use analgesic drugs.

Ages: 25 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-11-28 (Estimated); Study Completion 2021-12-28 (Estimated)

PRIMARY OUTCOMES:
Analgesia required | 24 hours
  time of first request for analgesia.

CONTACTS AND LOCATIONS:
Overall Officials: peter R Edward, MSc, Principal Investigator — specialist
Locations (1):
- South Egypt Cancer Institute, Asyut, Egypt